CLINICAL TRIAL: NCT04735341
Title: Prospective Post-market Data Collection for Ion Endoluminal System to Understand CT to Body Divergence
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-IonLR-001
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer; Pulmonary Nodule, Solitary
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with planned Ion Endoluminal Procedure with pulmonary nodule
  Interventions: Device: Ion Endoluminal System

INTERVENTIONS:
Device: Ion Endoluminal System — Ion Endoluminal Procedure for pulmonary nodule

SUMMARY:
The goal of this study is to collect post-market data for the Ion Endoluminal System to understand CT to body divergence.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older

  * Undergoing a lung biopsy procedure with Ion System
  * Have peripheral pulmonary lesion (5th bronchial generation or higher)
  * Willingness to participate as demonstrated by signing the informed consent

Exclusion Criteria:

* Unable to provide informed consent

  * Presence of bilateral nodules intended to be biopsied during procedure
  * The presence of medical conditions contraindicating general anesthesia or bronchoscopic biopsy
  * Vulnerable population (e.g., prisoners, mentally disabled)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who will undergo an Ion Endoluminal Procedure with a pulmonary nodule, 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Ion Catheter Shape | Intra-operative
  The collection of data relating to the Ion catheter shape

CONTACTS AND LOCATIONS:
Locations (1):
- FirstHealth of the Carolinas Moore Regional Hospital, Pinehurst, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No